CLINICAL TRIAL: NCT03203863
Title: Metabolic Syndrome in Adolescents. Associations With Endothelial Dysfunction and Early Programming Influences
Brief Title: Metabolic Syndrome in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor
Other Study IDs: 13-233; 1090594 (Other Grant/Funding Number: FONDECYT)
Record Dates: First submitted 2017-06-19; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Children; Cardiovascular; Risk Factors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Puente Alto, Chile, 2009-2011.: anthropometric measures of fatness
  Interventions: Diagnostic Test: anthropometric measures of fatness

INTERVENTIONS:
Diagnostic Test: anthropometric measures of fatness — The aim of this study was to determine the discrimination capacity for cardiovascular risk factors of BMI, fat mass (FM), waist circumference (WC), and waist to height ratio (WHtR) in a population of Chilean children from Puente Alto County. Additionally, new cutoff points were established and compared with those described by other authors

SUMMARY:
The purpose of this study was to cross-sectionally evaluate nutritional status and the metabolic syndrome in a sample of school-age children 10-15 years of age from 20 public schools in Santiago, Chile. In addition, the investigators retrospectively assessed the association of those variables with perinatal variables (birth weight, birth length, and gestational age at delivery).

DETAILED DESCRIPTION:
Subjects and methods Subjects The study was conducted in 2009-2011 in a cross-sectional way in 3,325 children attending 5th and 6th grade in 20 public schools of Santiago, Chile. All students were invited to participate in the study.

Anthropometry and other physical examinations Field measurements were performed by a nurse and a nutritionist. Height and weight were measured with children barefoot and lightly clothed using a stadiometer and a beam-scale Seca ®, with an accuracy of 50 g. The individual height and weight values were established by averaging three measurements of each parameter. BMI was calculated and expressed in percentiles and z-scores (13): z-scores were calculated according to Center for Disease Control-National Center of Statistics 2000. Nutritional status was classified according to BMI percentiles in the obese category as ≥ 95 (14). WC was measured with an inextensible tape on the upper lateral border of the right ilium in the mid-axillary line at the end of an exhalation (15) ; two measurements were averaged and the ≥ 90th percentile was used as cutoff value (16). The triceps and subscapular skin folds were measured with a Harpenden ® caliper using a standard technique (15); both were used to calculate the percentage of FM using Slaughter equations (17) previously validated in Chilean children (18, 19). Elevated FM was established as ≥ 42% for girls with 10-15 years old, ≥ 38% for boys with ≤ 12 years old, and 40% for boys with ≥ 13 years old (20).

A Critikon ® Dinamap Pro 100 BP monitor was used according to international norms and the averages of three measurements of systolic BP (SBP) were obtained and classified as abnormal using the ≥ 90 percentile of the same reference (21). A voluntary private self-report of pubertal status was requested by observation of standardized photos of breast development in girls and genitalia in boys including the presence of pubic hair (22). Maternal years of education were registered to estimate socio-economic level (23).

Blood samples Subjects were instructed to fast (water was allowed) for 12 hours prior to drawing of blood; non compliers were asked to return another day for the blood sampling. A single laboratory was used for all blood analyses at the Faculty of Medicine, Pontificia Universidad Católica de Chile.

Fasting venous blood samples were collected for determination of glucose (Gluco-quant method, Glucose / Hexokinase, Roche Diagnostics GmbH, Mannheim) and insulin (immunoassay direct luminometer chemotherapy, ADVIA Centaur ® XP, Bayer HealthCare LLC, Kyowa Medex Co. Japan); this method measures concentrations of insulin from 0.5 to 300 mUI / mL (sensitivity 0.5 mUI / mL) with a coefficient of variation of 3.48% and 6.17% for concentrations of 23.51 mUI / mL and 62.49 mUI / mL. respectively. Triglycerides and HDL-C were analyzed on the Modular Analytics P-800 platform (Roche Diagnostics GmbH, Mannheim, Germany).

ELIGIBILITY:
Inclusion Criteria:

The study was conducted in children attending 5th and 6th grade in all 20 public schools of the Municipality of Puente Alto, Santiago, Chile. All students were invited to participate in the study. Parents or their representatives signed an informed consent form and boys/girls an informed acceptance form.

Exclusion Criteria:

Subjects not signing the informed consent or acceptance forms were excluded from the study.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — A voluntary private self-report of pubertal status was requested by observation of standardized photos of breast development in girls and genitalia in boys including the presence of pubic hair (Tanner JM. Growth at adolescence. 2nd ed. Oxford: Blackwell Scientific Publications, 1962. ).
Study Population: Initially 5,614 students were eligible for the study (2,616 females and 2,998 males) but 2,289 students refused to participate (34.5% females and 47.4% males (p <0.001)). A total of 3,325 children and adolescents who presented a signed informed consent were included. No significant differences in age and years of maternal education were found between the study subjects and those who refused to participate.
Sampling Method: Non-Probability Sample
Enrollment: 3325 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2011-12-24 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Presence of metabolic syndrome | At recruitment
  Cardiovascular risk factors for children were used with the following cutoff points: SBP ≥ 90th percentile (20), low HDL-C ≤ 40 mg/dL; TG ≥ 110 mg/dL, and ≥ 90th percentiles of a Chilean HOMA standard for children, calculated according to sex and pubertal maturation, were used to classify insulin resistance (HOMA-IR).

IPD SHARING:
Plan to Share IPD: No